CLINICAL TRIAL: NCT01921478
Title: Retrospective, Multi-center, Observational Study of Daily Practice Patterns and Outcomes of the Management of Rheumatoid Arthritis Patients Without Documented Erosions Treated With RoACTEMRA in Belgium
Brief Title: A Retrospective, Observational Study of RoActemra/Actemra (Tocilizumab) in Clinical Practice in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25271
Record Dates: First submitted 2013-08-09; First posted 2013-08-13 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This retrospective, multi-centre, observational study will assess the daily practice patterns and outcomes of the management of rheumatoid arthritis in patients treated with RoActemra/Actemra (tocilizumab). No actual patient will be enrolled in this study; data will be collected from medical records.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >=18 years of age
* Diagnosed with rheumatoid arthritis and moderate to severe disease activity defined as a DAS28 >=5.1
* Inadequate responder to at least 2 non-biological DMARDs
* Absence of documented erosions at start of RoActemra/Actemra treatment
* Received RoActemra/Actemra treatment for at least 6 months
* Availability of data from at least the RoActemra/Actemra treatment initiation visit and the 6 months visit

Exclusion Criteria:

* Contraindications for treatment with RoActemra/Actemra

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective survey of medical records from patients with moderate to severe rheumatoid arthritis treated with RoActemra/Actemra (tocilizumab) who did not have documented erosions at the start of RoACTEMRA treatment .
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Joint erosion assessment in clinical practice | 6 months

SECONDARY OUTCOMES:
Disease Activity Score 28 | 6 months
C-reactive protein assessment | 6 months
Swollen joint counts | 6 months
Tender joint counts | 6 months
Erythrocyte Sedimentation Rate | 6 months
Evolution of the pattern of joint erosion | 6 months
Patient's global assessment of disease activity (Visual Analogue Scale) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Belgium (10):
  - Aalst
  - Antwerp
  - Bruges
  - Brussels
  - Ghent
  - Gilly
  - Seraing
  - Verviers
  - Westmalle
  - Wilrijk